CLINICAL TRIAL: NCT01451788
Title: Effectiveness Of Gelatin Matrix With Human Derived Thrombin On Blood Loss, Surgical Time, Hospital Stay And Complications In Adolescents Undergoing Spine Surgery For Adolescent Idiopathic Scoliosis: A Randomized Clinical Trial.
Brief Title: Effect of Human Thrombin With Gelatin Matrix on Perioperative Blood Loss in Scoliosis Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Tampere University Hospital (Other); Helsinki University Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TurkuUH
Record Dates: First submitted 2011-09-30; First posted 2011-10-14 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: RCT; Gelatin matrix; thrombin; idiopathic scoliosis; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional group (No Intervention): conventional blood saving methods (use of bone wax for cancellous bony bleeding; bipolar diathermy and epidural space packing for epidural venous bleeding)
- Floseal (Experimental): Gelatin matrix with human derived thrombin (Floseal) used in adolescents undergoing posterior spinal deformity surgery for adolescent idiopathic scoliosis (AIS)
  Interventions: Device: Gelatin matrix with human derived thrombin (Floseal, Baxter)

INTERVENTIONS:
Device: Gelatin matrix with human derived thrombin (Floseal, Baxter) — Floseal will be used to stop cancellous bone bleeding, pedicle channel bleeding or epidural space bleeding by injecting suitable amount of this matrix and irrigating it away after few minutes.
  Other Names: Floseal, Baxter
  Arms: Floseal

SUMMARY:
The Finnish Paediatric Orthopaedic Study Group will perform a prospective randomized, multicenter, clinical trial comparing Gelatin matrix with human derived thrombin (Floseal, Baxter) and without use of Floseal in adolescents undergoing posterior spinal deformity surgery for AIS (adolescent idiopathic scoliosis between 45 and 90 degrees) in Turku, Tampare and Helsinki Children's Hospitals. Sixty patients will be randomized into the intervention group receiving Floseal (n=30) and control group not receiving Floseal (n=30). Each University Hospital will treat 10 Floseal and 10 conventional treated scoliosis patients (block randomization). Both treatment groups will be allowed to use conventional blood saving methods.

DETAILED DESCRIPTION:
Background: Posterior spinal deformity surgery can be associated with major blood loss, especially from cancellous bone or epidural venous plexus. Products such as Gelatin Matrix with bovine derived thrombin (Floseal) can be used to prevent blood loss in adult patients undergoing spine surgery.

Aim: To document and compare effectiveness of Gelatin matrix with human derived thrombin with conventional blood loss control methods in adolescents undergoing posterior spinal deformity surgery for adolescent idiopathic scoliosis (AIS), who do not need vertebral column resection.

Methods: The Finnish Paediatric Orthopaedic Study Group will perform a prospective randomized, multicenter, clinical trial comparing Gelatin matrix with human derived thrombin (Floseal, Baxter) and without use of Floseal in adolescents undergoing posterior spinal deformity surgery for AIS (adolescent idiopathic scoliosis between 45 and 90 degrees) in Turku, Tampere and Helsinki Children's Hospitals. Sixty patients will be randomized into the intervention group receiving Floseal (n=30) and control group not receiving Floseal (n=30). Each University Hospital will treat 10 Floseal and 10 conventional treated scoliosis patients (block randomization). Both treatment groups will be allowed to use conventional blood saving methods.

Main outcome measures:

Blood loss during surgery (millilitres) Drain output during 24 hours (millilitres) Total blood loss (Blood loss during surgery + drain output, millitres) Used blood products (Red cell, frozen plasma, and thrombocyte units) Time of surgery Hospital stay Cost benefit analysis (blood product use, surgical time, hospital stay) Complications related to use of Floseal as a secondary outcome measure.

Primary Hypothesis and expected outcomes: Use of Floseal will reduce blood loss and surgical time in patients undergoing spine surgery for adolescent idiopathic scoliosis (Level-I evidence). Cost benefit analysis will most probably show that the use of Floseal is cost effective. E.g. the value of one allogenic Red Blood Cell unit is 400€. If no red blood cell units are needed instead of the usual three, the reduced blood product use alone will cover the extra costs of Floseal use. In addition, if no allogenic blood infusions are needed, the risk of infections will probably be significantly less. Reduced surgical time and shorter hospital stay may also be cost reducing findings in patients receiving Floseal.

Safety Aspects: Gelatin Matrix with human derived thrombin (Floseal, Baxter Biosurgery) is indicated for blood loss control in patients undergoing spine surgery when other methods are less effective.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be included if between 10 and 20 years of age, no contraindication for Floseal use, posterior scoliosis surgery using total pedicle screw technique for AIS with normal blood coagulation and normal whole spine magnetic resonance images except spinal deformity (AIS).

Exclusion Criteria:

* Need for anteroposterior surgery
* Need for vertebral column resection
* Smoking
* Diabetes mellitus
* Abnormalities in blood coagulation

Ages: 10 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Total perioperative blood loss | Surgery time (up to 8 hours) + first postoperative 24 hours
  Total blood loss during surgery + drain output, millilitres

SECONDARY OUTCOMES:
Used blood products | Surgery time (up to 8 hours) + first 24 hours postoperatively
  Red cell, frozen plasma, and thrombocyte units
Blood loss during surgery | up to 8 hours
  Blood loss during primary surgery, in millilitres
Time of surgery | up to 8 hours
  Time of surgery (hours, minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka J. Helenius, M.D., Ph.D., Study Director — Turku Children's Hospital, Turku University Central Hospital
Locations (3):
- Finland (3):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Central Hospital, Tampere
  - Turku Children's Hospital, Turku